CLINICAL TRIAL: NCT01915212
Title: Phase I Study of the Safety of a Replication-Defective Herpes Simplex Virus-2 Vaccine, HSV529, in Adults Aged 18 to 40 Years With or Without HSV Infection
Brief Title: Study of the Safety of a Particular Herpes Vaccine in Adults With or Without Herpes Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 130172; 13-I-0172
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2025-04-15

CONDITIONS: Healthy Volunteers
Keywords: Vaccination; Replication Defective; Genital Herpes; Safety; Immune Responses
MeSH Terms: conditions — Herpes Genitalis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HSV529 (Experimental): 1 x 107 pfu/dose of HSV529 in 10 mM L-histidine buffer containing 50 mM potassium glutamate, 160 mM sodium chloride, and 10% (w/v) sucrose
  Interventions: Biological: HSV529
- Placebo (Placebo Comparator): Sodium Chloride 0.9%
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: HSV529 — The vaccine was administered intramuscularly (deltoid muscle) as a 0.5 mL solution containing 1 x 10(7) plaque forming units on day 0, one month after the first dose (day 30) and then six months after the first dose (day 180).
  Arms: HSV529
Other: Placebo — Sodium Chloride 0.9%
  Arms: Placebo

SUMMARY:
Background:

- Herpes simplex virus type 2 (HSV-2) is a major cause of genital herpes. It can also cause serious infection in newborns and in people with weakened immune systems. It increases the risk of getting an HIV infection and of spreading HIV to someone else. Therefore, a vaccine that could prevent genital herpes could improve the general health of the world s population. Researchers want to study whether a new vaccine, HSV529, which may be used in the future to prevent herpes infections, is safe.

Objectives:

- To test whether a new herpes vaccine is safe.

Eligibility:

- Healthy adults 18 40 years old.

Design:

* Participants will have 3 vaccination visits, 7 follow-up visits, and 3 follow-up phone calls over 1 year.
* Each vaccination visit will last about 4 hours.
* Participants will be screened with a medical history and physical exam.
* Participants will have a blood sample taken.
* Participants will be given the vaccine or a placebo, by injection from a needle. They will be monitored for 30 minutes to check for any allergic reaction.
* Participants will be given a diary card to record any symptoms they may feel later.
* At follow-up visits, participants will give a blood sample and answer health questions.
* In the phone calls, participants will answer health questions.

DETAILED DESCRIPTION:
Herpes simplex virus 2 (HSV-2) causes genital herpes and increases the risk of acquisition and transmission of HIV. An HSV-2 vaccine is not available. We will study a replication-defective HSV-2 vaccine, HSV529, that is deleted for 2 essential viral proteins, that can infect, but not replicate in normal cells. The goals of the study are to determine (a) the safety of HSV529 vaccine in persons with or without HSV infection, and (b) the ability of the vaccine to elicit immune responses to HSV-2 including virus-specific antibodies and T cell responses to the virus. Three groups of 20 subjects each will be randomized and will receive 3 doses of HSV529 (15 subjects per group) or saline placebo injection (5 subjects per group). Each subject will be followed for 6 months after the last dose of vaccine. The 3 groups will be (a) subjects who were infected with HSV-2 in the past but may or may not have been infected with HSV-1 (HSV-1+/-/HSV-2+), (b) subjects who have been infected only with HSV-1 (HSV-1+/HSV-2-), and (c) subjects who have not been infected with HSV-1 or HSV-2 (HSV-1-/HSV-2-). Vaccine or placebo will be administered on Day 0 and approximately 1 month and 6 months after enrollment.

ELIGIBILITY:
* INCLUSION CRITERIA:

An individual must fulfill all of the following criteria in order to be eligible for trial enrollment:

1. Aged 18 to 40 years on the day of enrollment.
2. In good general health with absence of significant health problems as determined by medical history, physical examination, and laboratory screening performed during screening visits.
3. Subject will reside within a 60 mile or less radius from Bethesda, MD during the period of participation in the trial.
4. Hemoglobin, hematocrit, white blood cell count, platelet count, serum creatinine, and liver function (ALT, AST, alkaline phosphatase, total bilirubin) screening laboratory results do not fall into the range of values that are Grade 1 or greater as per the toxicity grading scale and IgG level greater than or equal to 600 mg/dl.
5. Females subjects must be of non-childbearing potential i.e. surgically sterilized (bilateral tubal ligation, hysterectomy) or, if of child-bearing potential and sexually active with a male partner, she must be willing to use a highly effective method of contraception (e.g., intrauterine device (IUD); oral contraceptives diaphragm or condom in combination with contraceptive foam, jelly or cream; Norplant, DepoProvera, contraceptive skin patch or cervical ring) for at least 30 days prior to vaccination and until 30 days after final vaccination or be in a monogamous relationship with a male partner who has undergone a vasectomy at least 6 months prior to first dose of study agent.
6. Willingness to attend all scheduled visits and able to comply with all trial procedures (e.g., blood draws, completion of diary cards, return for follow-up visits, accessible by phone or pager, able to self-sample for assessment of asymptomatic shedding of HSV, and not planning on moving from study area).
7. Negative HIV test result determined with an approved FDA-approved test. Confirmatory testing may be required based on the initial assay used and the result.
8. Subject is willing not to use antiviral therapy less than or equal to 2 days before and less than or equal to 3 days after each injection.
9. Subject is willing to forgo receipt of a licensed, live vaccine in the 30 days preceding each dose of vaccine or in the 30 days following each dose of vaccine. The inactivated flu vaccine can be used greater than or equal to 14 days before or greater than or equal to 14 days after administration of study vaccine, if this is felt to be necessary.
10. Persons who have close contact with infants or immunocompromised individuals agree to avoid such contact for 3 days after each injection.
11. Subject must be either HSV-1 IgG antibody positive or negative and HSV-2 IgG antibody positive, HSV-1 IgG antibody positive /HSV-2 IgG antibody negative, or HSV-1/HSV-2 IgG antibody negative as determined by an available commercial immunoassay.
12. Subject must be willing to allow storage of blood, swabs of skin or mucosa, biopsies of skin lesions, or, for female subjects, cervicovaginal secretions (if collected) for future research.

Participation of Women:

Contraception: The effects of HSV529 on the developing human fetus are unknown. For this reason, females subjects must be of non-childbearing potential i.e. either surgically sterilized (bilateral tubal ligation, hysterectomy) or, if of child-bearing potential and sexually active with a male partner, she must be willing to use a highly effective method of contraception (e.g., intrauterine device (IUD); oral contraceptives diaphragm or condom in combination with contraceptive foam, jelly or cream; Norplant, DepoProvera, contraceptive skin patch or cervical ring) for at least 30 days prior to vaccination and until 1 month after final vaccination or be in a monogamous relationship with a male partner who has undergone a vasectomy at least 6 months prior to first dose of study agent. Females must have a negative urine pregnancy test result prior to injection with HSV529 or placebo. During the course of the study, if a woman becomes pregnant or suspects she is pregnant, she should inform the study staff and her primary care physician immediately.

EXCLUSION CRITERIA:

Co-enrollment Guidelines: Co-enrollment in other trials is restricted, other than enrollment into observational studies or into the screening protocol. Study staff should be notified of co-enrollment as it may require the approval by the Principal Investigator.

An individual fulfilling any of the following criteria is to be excluded from trial enrollment:

1. Subject is pregnant or lactating OR planning to become pregnant timeframe that begins 30 days prior to the first vaccination and ends 30 days after the third vaccination.
2. Body Mass Index greater than 40.
3. Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the first trial vaccination or or planned participation during the study period up to 6 months after the last dose of vaccine or placebo. The non-interventional follow-up for an earlier study (e.g., long-term surveillance) will be allowed.
4. Severe active infection or serious HSV-2 related or unrelated medical conditions that, in the opinion of the investigator, would prevent study completion.
5. Subjects with 6 or more symptomatic recurrences of genital herpes disease within the year prior to Day 0.
6. A history of HSV infection of the eye (e.g., herpes simplex interstitial keratitis or uveitis).
7. A history of herpes gladiatorum, herpetic whitlow or eczema herpeticum.
8. A history of lesions caused by HSV on either arm.
9. A history of herpes-associated erythema multiforme.
10. A history of a clinically significant autoimmune disorder.
11. Known or suspected congenital or acquired immunodeficiency
12. Receipt of anti-cancer chemotherapy or radiation therapy within the preceding 6 months.
13. Subjects using corticosteroids (excluding topical, inhaled or nasal) or any immunomodulating drugs within 42 days prior to the first vaccination. An immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg prednisone equivalent per day for greater than or equal to 14 days.
14. Subjects without a spleen.
15. Subjects receiving immunoglobulin within the past 6 months or anticipated receipt of immunoglobulin during the 28 days following vaccination.
16. Bleeding disorder, or receipt of anticoagulants that, in the opinion of the Investigator, would interfere with the subject s participation in the trial.
17. Prior vaccination against herpes simplex virus.
18. Known allergy or intolerance to vaccine components [e.g., potassium glutamate (possible cross-reaction to monosodium glutamate), sucrose] or to a vaccine containing any of the same substances.
19. Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
20. Current alcohol abuse or drug abuse or addiction.
21. Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion.
22. Employee of the NIH or contractor working at the NIH, with direct involvement in the proposed study as well as family members (i.e. immediate, husband, wife and their children, adopted or natural) of the employee or of the investigators of this study.
23. Any condition that the PI thinks might compromise the person s ability to comply with the requirements of the study.

Justification for Exclusion of Women and Children:

Exclusion of Women:

* Pregnancy: Pregnant women are excluded from this study because the effects of HSV529 on the developing human fetus are unknown with the potential for teratogenic or abortifacient effects.
* Breast-feeding: Because there is an unknown but potential risk for adverse events in nursing infants secondary to vaccination of the mother with HSV529, breastfeeding should be discontinued if the mother will be vaccinated with HSV529.

Exclusion of Children:

Because there are insufficient data regarding dosing or adverse events available in adults to judge the potential risk in children, children are excluded from this study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2013-09-26 (Actual); Primary Completion 2017-03-06 (Actual); Study Completion 2017-03-06 (Actual)

PRIMARY OUTCOMES:
Unsolicited adverse events | After the first dose of vaccine to Day 360
  Safety
Solicited injection site and systemic reactions | Day 0 to Day 7 after each dose and up to day 360
  Safety

SECONDARY OUTCOMES:
Neutralizing antibody levels and T cell-mediated immune responses | After each dose and day 360
  Immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey I Cohen, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Da Costa XJ, Jones CA, Knipe DM. Immunization against genital herpes with a vaccine virus that has defects in productive and latent infection. Proc Natl Acad Sci U S A. 1999 Jun 8;96(12):6994-8. doi: 10.1073/pnas.96.12.6994. PMID 10359827
- [Background] Hoshino Y, Pesnicak L, Dowdell KC, Burbelo PD, Knipe DM, Straus SE, Cohen JI. Protection from herpes simplex virus (HSV)-2 infection with replication-defective HSV-2 or glycoprotein D2 vaccines in HSV-1-seropositive and HSV-1-seronegative guinea pigs. J Infect Dis. 2009 Oct 1;200(7):1088-95. doi: 10.1086/605645. PMID 19702506
- [Background] Da Costa X, Kramer MF, Zhu J, Brockman MA, Knipe DM. Construction, phenotypic analysis, and immunogenicity of a UL5/UL29 double deletion mutant of herpes simplex virus 2. J Virol. 2000 Sep;74(17):7963-71. doi: 10.1128/jvi.74.17.7963-7971.2000. PMID 10933704
- [Derived] Cheung F, Apps R, Dropulic L, Kotliarov Y, Chen J, Jordan T, Langweiler M, Candia J, Biancotto A, Han KL, Rachmaninoff N, Pietz H, Wang K, Tsang JS, Cohen JI. Sex and prior exposure jointly shape innate immune responses to a live herpesvirus vaccine. Elife. 2023 Jan 17;12:e80652. doi: 10.7554/eLife.80652. PMID 36648132
- [Derived] Dropulic LK, Oestreich MC, Pietz HL, Laing KJ, Hunsberger S, Lumbard K, Garabedian D, Turk SP, Chen A, Hornung RL, Seshadri C, Smith MT, Hosken NA, Phogat S, Chang LJ, Koelle DM, Wang K, Cohen JI. A Randomized, Double-Blinded, Placebo-Controlled, Phase 1 Study of a Replication-Defective Herpes Simplex Virus (HSV) Type 2 Vaccine, HSV529, in Adults With or Without HSV Infection. J Infect Dis. 2019 Aug 9;220(6):990-1000. doi: 10.1093/infdis/jiz225. PMID 31058977
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-I-0172.html